CLINICAL TRIAL: NCT00981136
Title: Single Incision Versus Standard Laparoscopic Appendectomy for Non-Perforated Appendicitis
Brief Title: Single Incision Laparoscopic Surgery (SILS) Versus Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09 07 133
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Appendicitis
Keywords: Appendicitis; Appendectomy; Children; Laparoscopic; SILS
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SILS (Active Comparator): Single Incision Laparoscopic Surgery (SILS) where a single incision in the umbilicus is all that is used to remove the appendix. The specific methods (staple/tie/port use/etc) will vary depending on surgeon.
  Interventions: Procedure: Single Incision Laparoscopic Appendectomy
- 3 port (Active Comparator): Standard laparoscopic appendectomy with 3 ports and intracorporeal stapling.
  Interventions: Procedure: 3 port laparoscopic appendectomy

INTERVENTIONS:
Procedure: Single Incision Laparoscopic Appendectomy — A single incision through the umbilicus to remove the appendix
  Other Names: SILS
  Arms: SILS
Procedure: 3 port laparoscopic appendectomy — Standard 3 port laparoscopic appendectomy with intracorporeal stapling
  Other Names: Laparoscopic Appendectomy
  Arms: 3 port

SUMMARY:
This is a prospective trial of single incision versus standard 3-port laparoscopic appendectomy.

The hypothesis is that there may a difference in wound infection rates, operative time, doses of analgesics post-operatively, and patient/parent perception of scars.

DETAILED DESCRIPTION:
This is a prospective, randomized clinical trial involving patients who present to the hospital with non-perforated appendicitis. We will offer enrollment to several institutions provided they receive institutional approval.

There are likely several parameters that will show small differences between groups, and this study will precisely quantify them to allow for adequate consultation from surgeons to families dealing with acute appendicitis. One theoretical concern over the SILS approach is that the exposure of the appendix to the wound could increase the rate of infectious complications; therefore, this is the primary outcome variable. The documented rate of infectious complications at our institution in patients with non-perforated appendicitis is 0.6%. An unacceptable and clinically relevant rise to 5% may curtail enthusiasm for the new technique. Using a power of 0.9 with an α of 0.05, the sample size is 360 total patients or 180 in each arm.

After the procedure, both groups will be managed in the same manner per routine care. They will be discharged when tolerating a regular diet and their pain is well-controlled on oral pain medication. Cosmetic scores will be obtained at 6 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years
* Non-perforated appendicitis

Exclusion Criteria:

* Perforated appendicitis as identified as a hole in the appendix for fecalith in the abdomen

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Post-operative infection | 6 weeks

SECONDARY OUTCOMES:
Doses of analgesic | 3 days
Operative time | 1 day
Cosmetic scores | 6 months
Length of Hospitalization | 1 week
Surgeon perception of difficulty | 1 day
Hospital/operative charges | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Shawn d St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Derived] St Peter SD, Shah SR, Adibe OO, Sharp SW, Reading B, Cully B, Holcomb GW 3rd, Rivard DC. Saline vs Tissue Plasminogen Activator Irrigations after Drain Placement for Appendicitis-Associated Abscess: A Prospective Randomized Trial. J Am Coll Surg. 2015 Aug;221(2):390-6. doi: 10.1016/j.jamcollsurg.2015.03.043. Epub 2015 Mar 30. PMID 26141467
- [Derived] St Peter SD, Adibe OO, Iqbal CW, Fike FB, Sharp SW, Juang D, Lanning D, Murphy JP, Andrews WS, Sharp RJ, Snyder CL, Holcomb GW, Ostlie DJ. Irrigation versus suction alone during laparoscopic appendectomy for perforated appendicitis: a prospective randomized trial. Ann Surg. 2012 Oct;256(4):581-5. doi: 10.1097/SLA.0b013e31826a91e5. PMID 22964730
- [Derived] St Peter SD, Adibe OO, Juang D, Sharp SW, Garey CL, Laituri CA, Murphy JP, Andrews WS, Sharp RJ, Snyder CL, Holcomb GW 3rd, Ostlie DJ. Single incision versus standard 3-port laparoscopic appendectomy: a prospective randomized trial. Ann Surg. 2011 Oct;254(4):586-90. doi: 10.1097/SLA.0b013e31823003b5. PMID 21946218